CLINICAL TRIAL: NCT06769945
Title: The Effect of Nursing Care Based on Kolcaba's Comfort Theory on the Comfort Levels of Patients Undergoing Open Heart Valve Surgery
Brief Title: Kolcaba's Comfort Theory on the Comfort Levels of Patients Undergoing Open Heart Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Ozkan Sir, lecturer, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ataturk Unıversity; TDK-2024-14325 (Other: Ataturk Unıversıty)
Record Dates: First submitted 2024-12-13; First posted 2025-01-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Surgery (Cardiac)
MeSH Terms: interventions — Patient Education as Topic; Pain Management

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Patients in the experimental group will receive nursing care based on Kolcaba's Comfort Theory during their stay in the cardiovascular surgery service. After determining the comfort-oriented care needs of the patients, the General Comfort Scale will be used and individualised nursing care plans will be created in line with these needs. According to Kolcaba, standard comfort interventions and comfort interventions provided by coaching will be applied.
  Interventions: Behavioral: Nursing Care Based on Kolcaba's Comfort Theory
- Control (No Intervention): Control group patients will receive routine nursing care in the ward environment.

INTERVENTIONS:
Behavioral: Nursing Care Based on Kolcaba's Comfort Theory — In practice, patient education, pain management, emotional support, appropriate environmental arrangements and individualised care come to the fore. Studies show that with this approach, patients' physical comfort increases, anxiety levels decrease and overall satisfaction improves. It is stated that nursing care based on Kolcaba's theory offers an effective model to improve the quality of life of postoperative patients.
  Other Names: In practice, patient education, pain management, emotional support, appropriate environmental arrangements and individualised care come to the fore. Studies show that with this approach, patients' phy
  Arms: experimental

SUMMARY:
It is planned to determine the effect of comfort theory-based nursing care on the comfort and pain levels of patients undergoing open heart valve surgery.

* Does nursing care based on comfort theory reduce the comfort of patients undergoing open heart valve surgery?
* Does nursing care based on comfort theory reduce the pain level of patients undergoing open heart valve surgery?
* Does nursing care based on comfort theory increase the comfort level of patients undergoing open heart valve surgery?
* Does nursing care based on comfort theory increase the pain level of patients undergoing open heart valve surgery?

DETAILED DESCRIPTION:
Comfort is defined as "an expected result with a complex structure within the physical, psychological, social and environmental integrity of helping the individual with his/her needs, providing peace of mind and being able to overcome problems." In his theory, Kolcaba defined comfort as "an expected result with a complex structure within the physical, psychospiritual, social and environmental integrity of helping the individual with his needs, providing peace of mind and overcoming problems. This situation affects recovery and discharge times. Studies indicate that comfort is one of the most important factors affecting the speed of recovery. The sample size of the study was determined using power analysis. As a result of the Power analysis (G*Power 3.1.9.4); when the effect size was taken as Cohen's d: 0.95, the number of samples determined for a confidence interval of 95%, a power of 95%, and a margin of error of 0.05 was determined as a total of 50 patients, with a minimum of 25 patients for each group (Experimental and Control). Considering the block randomization distributions, the study was completed with 56 patients.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being 18 years of age or older,
* Being open to communication,
* Not having any obstacle in terms of consciousness and sensory organs,
* Being in the cardiovascular surgery service clinic

Exclusion Criteria:

* Hearing and/or visual loss
* Leaving the study voluntarily
* Patients transferred from the ward environment back to the intensive care environment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
comfort | To be filled in at 0th and 72nd hours of nursing care.
  General Comfort Scale:The highest total score that can be obtained from the scale is 192, and the lowest total score is 48. Low comfort represents one point, and high comfort represents four points.
  Time frame: To be filled in at 0th and 72nd hours of nursing care.
VAS (Visual Analog Scale) Pain | To be filled in at 0th and 72nd hours of nursing care
  VAS ( Visual analog scale) On a line with '0' on one end and '10' on the other, patients will be asked to choose, explaining that 0 means no symptoms and 10 means the most severe symptoms. A high score here indicates that the patient has high pain during the treatment and care process.
  Time frame: To be filled in at 0th and 72nd hours of nursing care

CONTACTS AND LOCATIONS:
Locations (1):
- VAN, Erzurum, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No